CLINICAL TRIAL: NCT04606966
Title: Physiological Mechanisms of Action Relating to Immediate and Long-term Therapeutic Horseback Riding Intervention Effects in a Psychiatric Population of Youth With Autism Spectrum Disorder
Brief Title: Physiological Mechanisms of Therapeutic Horseback Riding Intervention Effects in a Psychiatric Population of ASD Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Maine Health/Spring Harbor Hospital (Unknown); Riding To The Top Therapeutic Riding Center (Unknown); Hearts and Horses Therapeutic Riding Center (Unknown); Salimetrics, LLC (Unknown); Baylor University (Other); University of Pittsburgh (Other); Colorado State University (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1962; 1R01HD097693-01A1 (NIH)
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder; Mental Disorders
Keywords: human-animal intervention; physiology; mechanisms of action; children; adolescents; emotion regulation; cortisol; heart rate; electrodermal activity
MeSH Terms: conditions — Autism Spectrum Disorder; Mental Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial assigned to one of 3 groups:
  Therapeutic Horseback Riding group Barn Activity group (no-horse control) Waitlist Hybrid group
Who Masked: Outcomes Assessor
Masking Description: Speech therapist evaluator will be blinded to participants' intervention condition assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Therapeutic Horseback Riding (Experimental): This Arm is a 10 week one hour small group (2-4 participants) led by a THR instructor. The group will include a 45-minute mounted activity to learn horsemanship skills as outlined in the study's THR manual, . Group times will be between 1:00-5:00 PM to collect salivary cortisol. Weekly, participants will follow a consistent routine of wearing both their electro dermal activity and heart rate monitoring devices, sit at a group art table before class, after this, study personnel will instruct participants to place the 10cm long foam swab rod under their tongue for one minute while watching a 1-minute timer. Participants will then don their riding helmets and enter the riding arena. Each week after conclusion of the THR intervention, participants will again sit with their group at an art table for 5 minutes followed by doing another saliva sample.
  Interventions: Other: Therapeutic Horseback Riding
- Barn Activity (Active Comparator): This Arm is a 10 week one hour small group (2-4 participants) led by a THR instructor and co-led by a mental health or Occupational therapy provider. Participants will have one assigned volunteer and will have no physical contact with horses at the riding center, just view horses from a distance. There will be a life-sized stuffed toy horse for hands-on learning related to the weekly topic per the BA study manual. Group times will be between 1:00-5:00 PM to collect salivary cortisol. Weekly, participants will follow a consistent routine of wearing both their electro dermal activity and heart rate monitoring devices, sit at a group art table before class, after this, study personnel will instruct participants to place the 10cm long foam swab rod under their tongue for one minute while watching a 1-minute timer. Each week after conclusion of the BA intervention, participants will again sit with their group at an art table for 5 minutes followed by doing another saliva sample.
  Interventions: Other: Barn Activity
- Waitlist (No Intervention): Those assigned to the waitlist group will not have any horse-related intervention during a 10-week waiting period. Following this waiting period and the completion of post assessments, participants in this condition will begin a Hybrid group (see Hybrid Arm)
- Hybrid (Experimental): Participants completing the Wait list Arm and post assessments, will begin a Hybrid group between 1:00-5:00 PM. The group consists of a 5- week 1 -hour BA small group (2-4 participants) led by a THR instructor and co-led by a mental health counselor or OT. Participants will have one assigned volunteer and have no physical contact with horses at the riding center, just view horses at a distance. There will be a life-sized stuffed horse for hands-on learning weekly topics per BA study manual. Group. Then, participants will complete 5-weeks of Therapeutic Horseback Riding small group (2-4 participants) led by a THR instructor. The group will include a 45-minute mounted activity to learn horsemanship skills followed by a 15-minute unmounted horse grooming and tacking activity per THR manual. Participants will have an assigned horse and volunteer(s).
  Interventions: Other: Hybrid

INTERVENTIONS:
Other: Therapeutic Horseback Riding — Horse therapy
  Other Names: Equine Assisted Activity
  Arms: Therapeutic Horseback Riding
Other: Barn Activity — Horsemanship group
  Other Names: No Horse control
  Arms: Barn Activity
Other: Hybrid — Ground and riding activities
  Other Names: Equine Assisted Activity
  Arms: Hybrid

SUMMARY:
This randomized control trial (RCT) seeks to assess the mechanisms underlying Therapeutic Horseback Riding's (THR) previously observed significant positive effects on ASD youth, particularly those with co-occurring psychiatric disorders, and to refine information on the durability, dose and sub-population effects of the intervention.

DETAILED DESCRIPTION:
This randomized control trial (RCT) will test the hypothesis that physiological response patterns of salivary cortisol, cardiovascular, and electrodermal activity account for our previously observed significant outcomes (i.e., reduced irritability and hyperactivity, and improved social and communication), and additional outcomes (emotion regulation caregiver quality of life and crisis mental health care usage), in youth ages 6-16 yrs. with ASD and co-occurring psychiatric diagnoses randomized to a 10-week manualized THR intervention compared to a no-horse Barn Activity (BA) control (Aim 1). We will evaluate the durability of Aim 1 outcomes in the THR group compared to the BA control group six-months after the intervention period (Aim 2). Finally, we will explore dose and sub-population effects of THR and BA interventions by comparing effect size differences in THR and BA groups to (a) a 10-week wait-list control group; (b) a Hybrid intervention group (five weeks BA followed by five weeks THR); and (c) a subsample of the THR study population randomized following psychiatric hospitalization (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* documented ASD diagnosis and a co-occurring psychiatric disorder
* ABC Irritability subscale score ≥8
* Leiter-III Nonverbal IQ ≥ 40
* meet Symptom Criterion score (minimum number of symptoms necessary for a DSM-V (mood, anxiety, or ADHD diagnosis) on CASI-5)
* meet ASD cut-offs on the SCQ (≥ 11) and on ADOS-2
* Only one child with ASD per family to maintain independent observations
* a consistent caregiver (i.e., parent or legal guardian) to complete study outcome measures

Exclusion Criteria:

* medical or behavioral issues that prevent participation
* ward of the state
* judged during riding center screen to have significant riding experience
* smoking or regular use of oral, inhaled, or topical steroids on a regular basis, factors known to affect cortisol levels
* Participants weighing 200 pounds or greater will be excluded due to the riding center's safety policies
* Participants will not be allowed to begin baseline assessments until at least six months have passed from the time they last engaged in mounted EAAT, given pilot evidence for the six-month maintenance of THR effects.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist-Community (ABC-C) | Baseline, week 10, 6 months
  58-item symptom presence and severity (0-3, not a problem to severe problem) checklist of problem behaviors of children and adults with developmental disabilities in community settings. The 58 items resolve into five subscales: (1) Irritability, Agitation, (2) Lethargy, Social Withdrawal, (3) Stereotypic Behavior, (4) Hyperactivity, and (5) Inappropriate Speech.Irritability and Hyperactivity behaviors
Change in Social Responsiveness Scale™, Second Edition | Baseline, week 10, 6 months
  social awareness, social cognition, social communication, social motivation, autistic mannerisms. Results in a T-score that indicates severity level ranges.
Change in Emotion Dysregulation Inventory (EDI) | Baseline, week 10, 6 months
  24 -item Reactivity behaviors of intense, rapidly escalating, sustained, and poorly regulated negative emotional reactions, and 6-item Dysphoria behaviors of minimal positive affect and motivation, and the presence of nervousness and sadness.Both the Dysphoria Scale and Reactivity Short Form have IRT-based theta scores, which have a mean of 0 and SD of 1, and provide superior discriminative ability to raw scores.
Change in World Health Organization's Quality of Life Instrument (WHOQOL-BREF) | Baseline, week 10, 6 months
  Quality of life for caregiver
Change in Systematic Analysis of Language Transcripts (SALT) | Baseline, week 10, 6 months
  Expressive Language Sample
Change in Crisis Mental Health Care Usage Survey | Baseline, week 10, 6 months
  crisis mental health care usage

OTHER OUTCOMES:
Change in Salivary Cortisol | Baseline, Midpoint Intervention (about Week 5), Week 10
  Mediator
Change in Electrodermal Activity | Baseline, Midpoint Intervention (about Week 5), Week 10
  Change in skin conductance will be reported. Electrodes will be attached to the underside of the wrist of their non-dominant hand to record electrodermal activity (EDA). EDA measures individual differences in endocrine sweat gland activity.
Change in Heart Rate/Heart Rate Variability | Baseline, Midpoint Intervention (about Week 5), Week 10
  Mediator

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Gabriels, Psy.D., Principal Investigator — University of Colorado Anzchutz Medical Campus
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Maine Health, Portland, Maine

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT04606966/Prot_001.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT04606966/ICF_000.pdf